CLINICAL TRIAL: NCT06119139
Title: Anesthetic Efficacy of 1.8 ml Compared to 3.6 ml of Articaine Buccal Infiltration in Mandibular Molars With Symptomatic Irreversible Pulpitis: A Randomized Clinical Trial
Brief Title: Anesthetic Efficacy of 1.8 ml Versus 3.6 ml of 4% Articaine Buccal Infiltration
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hebatullah Moheb Ibrahim, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CU-Endo.23.10.23
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Symptomatic Irreversible Pulpitis
MeSH Terms: interventions — Carticaine

STUDY DESIGN:
Intervention Model Description: Parallel, randomized, clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1.8 ml 4% articaine buccal infiltration. (Active Comparator)
  Interventions: Drug: 1.8 ml 4% Articaine hydrochloride
- 3.6 ml 4% articaine buccal infiltration (Experimental)
  Interventions: Drug: 3.6 ml 4% Articaine hydrochloride

INTERVENTIONS:
Drug: 3.6 ml 4% Articaine hydrochloride — 3.6 ml 4% articaine buccal infiltration
  Arms: 3.6 ml 4% articaine buccal infiltration
Drug: 1.8 ml 4% Articaine hydrochloride — 1.8 ml 4% articaine buccal infiltration
  Arms: 1.8 ml 4% articaine buccal infiltration.

SUMMARY:
The aim of the study is to compare the anesthetic efficacy and need for supplemental anesthesia of 1.8 ml compared to 3.6 ml of 4% articaine buccal infiltration in mandibular molars with symptomatic irreversible pulpitis.

DETAILED DESCRIPTION:
Patients with moderate-to-severe pain due to symptomatic irreversible pulpitis will be included. Patients will be randomly assigned into two groups to receive either 1.8 ml 4% articaine buccal infiltration or 3.6. ml 4% articaine buccal infiltration before single visit root canal treatments. Intraoperative pain will be assessed using an 11-point numerical rating scale (NRS) so that anesthetic success will be defined as no to mild intraoperative pain. The need for supplemental anesthesia will also be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy patients who are categorized as I or II according to The American Society of Anesthesiologists (ASA class I or II).
2. No sex predilection
3. Patients with symptomatic irreversible pulpitis
4. Patient with the ability to understand and use pain scales.
5. Patients who accept to enroll in the study.

Exclusion Criteria:

1. Patients' allergies to any of the drugs or materials used in the study.
2. Pregnant and lactating females.
3. Patients taking analgesics in the last 6-8 hours.
4. Patients having more than one symptomatic tooth in the same quadrant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Anesthetic success | During the procedure
  Will be measured by 11-point numerical rating scale NRS. The success will be defined as no or mild pain (NRS 0 or less than 3) and the failure will be defined as moderate to severe pain (NRS more than 3).

SECONDARY OUTCOMES:
Need for supplemental anesthesia | During the procedure
  Whether the patient requires supplemental anesthesia or not. It will be recorded by the questionnaire (yes or no).

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Poorni S, Veniashok B, Senthilkumar AD, Indira R, Ramachandran S. Anesthetic efficacy of four percent articaine for pulpal anesthesia by using inferior alveolar nerve block and buccal infiltration techniques in patients with irreversible pulpitis: a prospective randomized double-blind clinical trial. J Endod. 2011 Dec;37(12):1603-7. doi: 10.1016/j.joen.2011.09.009. PMID 22099890
- [Background] Abazarpoor R, Parirokh M, Nakhaee N, Abbott PV. A Comparison of Different Volumes of Articaine for Inferior Alveolar Nerve Block for Molar Teeth with Symptomatic Irreversible Pulpitis. J Endod. 2015 Sep;41(9):1408-11. doi: 10.1016/j.joen.2015.05.015. Epub 2015 Jul 3. PMID 26149210
- [Background] Monteiro MR, Groppo FC, Haiter-Neto F, Volpato MC, Almeida JF. 4% articaine buccal infiltration versus 2% lidocaine inferior alveolar nerve block for emergency root canal treatment in mandibular molars with irreversible pulpits: a randomized clinical study. Int Endod J. 2015 Feb;48(2):145-52. doi: 10.1111/iej.12293. Epub 2014 May 22. PMID 24702239